CLINICAL TRIAL: NCT05485961
Title: A Phase 2b / 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Combined Dose-Finding and Cardiovascular Outcome Study to Investigate the Efficacy and Safety of CSL300 (Clazakizumab) in Subjects With End Stage Kidney Disease Undergoing Dialysis
Brief Title: Combined Dose-Finding and CV Outcomes Study With CSL300 (Clazakizumab) in Adult Subjects With ESKD Undergoing Dialysis
Acronym: POSIBIL6ESKD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CSL300_2301; 2022-500273-14-00 (Other: EU CT)
Record Dates: First submitted 2022-07-29; First posted 2022-08-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-08

CONDITIONS: Atherosclerotic Cardiovascular Disease; End Stage Kidney Disease; Atherosclerotic Cardiovascular Disease in Patients With ESKD
Keywords: End Stage Kidney Disease (ESKD); Myocardial infarction (MI); Atherosclerotic cardiovascular disease (ASCVD); Coronary artery disease; Peripheral artery disease; Diabetes
MeSH Terms: conditions — Atherosclerosis; Kidney Failure, Chronic; Myocardial Infarction; Coronary Artery Disease; Peripheral Arterial Disease; Diabetes Mellitus | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CSL300 (low dose)(Phase 2b) (Experimental): Intravenous (IV) administration
  Interventions: Drug: CSL300
- CSL300 (medium dose)(Phase 2b) (Experimental): IV administration
  Interventions: Drug: CSL300
- CSL300 (high dose)(Phase 2b) (Experimental): IV administration
  Interventions: Drug: CSL300
- Placebo (Phase 2b) (Placebo Comparator): IV administration
  Interventions: Drug: Placebo
- CSL300 (Phase 3) (Experimental): IV administration
  Interventions: Drug: CSL300
- Placebo (Phase 3) (Placebo Comparator): IV administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSL300 — IV administration
  Other Names: Clazakizumab
  Arms: CSL300 (Phase 3); CSL300 (high dose)(Phase 2b); CSL300 (low dose)(Phase 2b); CSL300 (medium dose)(Phase 2b)
Drug: Placebo — Matching the excipient content and concentration of the CSL300 product, minus the active ingredient.
  Arms: Placebo (Phase 2b); Placebo (Phase 3)

SUMMARY:
This is a 2-part (phase 2b/3) prospective, interventional, multicenter, randomized, double-blind, placebo-controlled study. Part 1 (phase 2b) is a dose-finding study for CSL300 vs placebo. Part 2 (phase 3) aims to assess the efficacy of CSL300 on cardiovascular (CV) outcomes and safety in subjects with systemic inflammation and either atherosclerotic cardiovascular disease (ASCVD) or diabetes with end stage kidney disease (ESKD) undergoing maintenance dialysis.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female at least 18 years of age
* - A diagnosis of ESKD undergoing maintenance dialysis for at least 12 weeks
* - Serum hs-CRP ≥ 2.0 mg/L
* - A diagnosis of diabetes mellitus OR ASCVD

Exclusion Criteria:

* - Subjects who participated in Part 1 (phase 2b) are not eligible to participate in Part 2 (phase 3)
* - Concomitant use of systemic immunosuppressant drugs
* - Abnormal LFTs
* - Any life-threatening disease expected to result in death within 12 months
* - A history of GI perforation, inflammatory bowel disease (except fully excised ulcerative colitis), or peptic ulcer disease
* -Clinically significant active infection or history of opportunistic or invasive fungal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2310 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the log scale in high-sensitivity C-reactive protein (hs-CRP)(Phase 2b) | Baseline and up to 12 weeks
Time to first occurrence of CV death or myocardial infarction (MI) (Phase 3) | Approximately 5 years

SECONDARY OUTCOMES:
Percent of participants achieving hs-CRP less than (<) 2.0 milligram per Liter (mg/L) (Phase 2b) | Week 12
Change from baseline in log-transformed hs-CRP (Phase 2b) | Baseline and up to 24 weeks
Mean change from Baseline in serum amyloid A (SAA) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in secretory phospholipase A2 (sPLA2) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in fibrinogen (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in plasminogen activator inhibitor -1 (PAI-1) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in lipoprotein (Lp) (a) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in albumin (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in Hepcidin (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in hemoglobin (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in erythropoiesis-stimulating agents (ESA) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in erythropoietin-resistance index (ERI) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in iron (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in total iron binding capacity (TIBC) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in transferrin saturation (TSAT) (Phase 2b) | Baseline and up to 12 weeks
Mean change from Baseline in ferritin (Phase 2b) | Baseline and up to 12 weeks
Area under the plasma concentration versus time curve (AUC) for CSL300 (Phase 2b) | Up to 24 weeks
Peak Plasma Concentration (Cmax) for CSL300 (Phase 2b) | Up to 24 weeks
Trough Plasma Concentration (Ctrough) for CSL300 (Phase 2b) | Up to 24 weeks
Time to Maximum Plasma Concentration (Tmax) for CSL300 (Phase 2b) | Up to 24 weeks
Percent of participants with adverse events (AE), serious AE (SAE), including adverse events of special interest (AESIs) (Phase 2b) | Up to 32 weeks
Mean change from Baseline in white blood cell (WBC) (Phase 2b) | Up to 12 weeks
Mean change from Baseline in neutrophils (Phase 2b) | Up to 12 weeks
Mean change from Baseline in platelets (Phase 2b) | Up to 12 weeks
Mean change from Baseline in aspartate aminotransferase (AST) (Phase 2b) | Up to 12 weeks
Mean change from Baseline in alanine aminotransferase (ALT) (Phase 2b) | Up to 12 weeks
Mean change from Baseline in total bilirubin (Phase 2b) | Up to 12 weeks
Mean change from Baseline in lipid panel (Phase 2b) | Up to 12 weeks
  Lipid panel consists of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), triglyceride.
Titer of confirmed antibodies specific to CSL300 (Phase 2b) | Up to 12 weeks
Time to first occurrence of all-cause death or MI (Phase 3) | Approximately 5 years
Time to first occurrence of CV death, MI, or ischemic stroke (Phase 3) | Approximately 5 years
Time to first occurrence of CV death (Phase 3) | Approximately 5 years
Time to first occurrence of CV death, MI or major adverse limb event (Phase 3) | Approximately 5 years
Time to first occurrence of all-cause death (Phase 3) | Approximately 5 years
Time to first occurrence of CV death, MI, or hospitalization for heart failure (HF) (Phase 3) | Approximately 5 years
Total number of CV hospitalizations (Phase 3) | Approximately 5 years
Total number of HF hospitalizations and urgent visits (Phase 3) | Approximately 5 years
Total number of hospitalizations (Phase 3) | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring LLC
Locations (413):
- United States (156):
  - Nephrology of North Alabama, Decatur, Alabama
  - 84000149 - Nephrology Consultants, LLC, Huntsville, Alabama
  - 84000340 - DaVita Clinical Research Montgomery, Montgomery, Alabama
  - 84000552 - AKDHC Medical, Glendale, Arizona
  - 84000178 - Kidney Disease Medical Group, Glendale, Arizona
  - 84000231 - AKDHC Medical, Phoenix, Arizona
  - 84000286 - AKDHC Medical, Tucson, Arizona
  - 84000622 - Southern Arizona VA Health Care System, Tucson, Arizona
  - 84000145 - National Institute of Clinical Research, Bakersfield, California
  - 84000151 - National Institute of Clinical Research, Bakersfield, California
  - 84000277 - Amicis Research Center, Beverly Hills, California
  - 84000241 - California Institute of Renal Research, Chula Vista, California
  - The Medical Research Group, Inc., Fresno, California
  - 84000462 - Davita Fullerton Dialysis Center, Fullerton, California
  - 84000574 - National Institute of Clinical Research, Inc., Fullerton, California
  - 84000464 - St. Jude Medical Center, Garden Grove, California
  - 84000573 - National Institute of Clinical Research, Inc., Garden Grove, California
  - 84000152 - National Institute of Clinical Research, Garden Grove, California
  - 84000531 - Sherman Medical Group, Inc, Glendale, California
  - 84000230 - Kidney Disease Medical Group, Glendale, California
  - 84000379 - Renal Consultants Medical Group, Granada Hills, California
  - 84000631 - Balboa Research, La Jolla, California
  - 84000221 - California Institute of Renal Research, La Mesa, California
  - 84000235 - California Institute of Renal Research, La Mesa, California
  - 84000198 - Southern California Medical Research Center, La Palma, California
  - 84000467 - Southern California Medical Research Center, La Palma, California
  - 84000329 - Academic Medical Research Institute, Los Angeles, California
  - 84000439 - National Institute of Clinical Research, Inc., Los Angeles, California
  - 84000158 - DaVita Carabello Dialysis Center, Los Angeles, California
  - 84000175 - Renal Medical Associates/NARI, Lynwood, California
  - 84000279 - Amicis Research Center, Northridge, California
  - 84000533 - FORMAT Medical Research, Oxnard, California
  - 84000331 - Van Buren Dialysis Center, Riverside, California
  - 84000228 - National Nephrology Alliance Research - Riverside, Riverside, California
  - 84000492 - Central Coast Nephrology Medical Corp, Salinas, California
  - 84000238 - California Institute of Renal Research, San Diego, California
  - 84000143 - California Institute of Renal Research, San Diego, California
  - 84000330 - North America Research Institute, San Dimas, California
  - 84000341 - North America Research Institute, San Dimas, California
  - 84000281 - Satellite Healthcare, San Jose, California
  - 84000440 - Nephrology Educational Services, Tarzana, California
  - 84000536 - Valiance Clinical Research, Tarzana, California
  - 84000278 - Amicis Research Center, Vacaville, California
  - 84000323 - National Institute of Clinical Research, Inc, Victorville, California
  - 84000174 - DaVita Vista Del Sol Dialysis, Victorville, California
  - 84000589 - Western Nephrology, Arvada, Colorado
  - 84000454 - Kidney Associates of Colorado, P.C., Denver, Colorado
  - 84000223 - Colorado Kidney Care, Denver, Colorado
  - 84000176 - Greater Hartford Nephrology, LLC, Bloomfield, Connecticut
  - 84000173 - Nephrology and Hypertension Associates PC, Middlebury, Connecticut
  - 84000494 - Nephrology Associates (Delaware), Newark, Delaware
  - 84000441 - Boca Raton Regional - Research Physicians Network Alliance, Boca Raton, Florida
  - 84000779 - Nova Clinical Research, LLC, Bradenton, Florida
  - 84000661 - Access Research Institute, Brooksville, Florida
  - 84000193 - Horizon Research Group LLC, Coral Gables, Florida
  - 84000443 - South Florida Nephrology Group, PA, Coral Springs, Florida
  - 84000597 - Family First Medical Research Center, Hialeah Gardens, Florida
  - 84000650 - Advanced Medical Research Group, Hollywood, Florida
  - 84000406 - Elixia Pines, Hollywood, Florida
  - 84000140 -South Florida Research Institute, Lauderdale Lakes, Florida
  - 84000599 - South Florida Research Organization LLC, Medley, Florida
  - Aviva Health Sciences, Miami, Florida
  - 84000495 - Total Research Group, LLC, Miami, Florida
  - 84000663 - Iconic Clinical Research Center, Miami, Florida
  - 84000362 - Kidney and Hypertension Specialists of Miami, Miami, Florida
  - 84000182 - Nephrology Associates of South Miami, Miami, Florida
  - 84000527 - Floridian Clinical Research, Miami Lakes, Florida
  - 84000400 - Elixia Central Florida, Orlando, Florida
  - Infigo Clinical Research LLC, Sanford, Florida
  - 84000139 - Genesis Clinical Research, Tampa, Florida
  - 84000532 - Florida Kidney Specialists, Temple Terrace, Florida
  - 84000426 - Florida Premier Research Institute, Winter Park, Florida
  - 84000366 - Southwest Georgia Nephrology Clinic, Albany, Georgia
  - 84000326 - Coastal Medical Research, LLC, Brunswick, Georgia
  - 84000157 - Renal Associates LLC, Columbus, Georgia
  - National Clinical Trials, Cordele, Georgia
  - 84000327 - American Clinical Trials, Douglasville, Georgia
  - 84000582 - Georgia Nephrology, Lawrenceville, Georgia
  - 84000194 - Atekha Nephrology Clinic LLC, Statesboro, Georgia
  - 84000528 - NANI Research, Fort Wayne, Indiana
  - 84000453 - Nephrology Physician's LLC, Mishawaka, Indiana
  - 84000534 - Dunes Clinical Research LLC, Sioux City, Iowa
  - 84000374 - Kansas Nephrology Physicians, PA, Wichita, Kansas
  - 84000554 - Nephrology Associates of Kentuckiana, PSC, Louisville, Kentucky
  - 84000550 - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - 84000220 - Massachusetts General Hospital, Boston, Massachusetts
  - 84000465 - Paragon Health, Inc, Kalamazoo, Michigan
  - 84000408 - Michigan Kidney Consultants, PC, Pontiac, Michigan
  - 84000171 - St. Clair Nephrology Research, Roseville, Michigan
  - 84000237 - Center for Advanced Kidney Research, PLC, Saint Clair Shores, Michigan
  - 84000146 - DCR Edina, Minneapolis, Minnesota
  - 84000338 - DCR Edina, Minneapolis, Minnesota
  - 84000225 - Southwest Mississippi Nephrology PLLC, Brookhaven, Mississippi
  - 84000153 - Nephrology Associates, PC, Columbus, Mississippi
  - 84000144 - Nephrology and Hypertension Associates Ltd, Tupelo, Mississippi
  - 84000147 - Clinical Research Consultants, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - 84000377 - DCI-Rockhill, Kansas City, Missouri
  - 84000328 - GSR Enterprises, Inc., Lincoln, Nebraska
  - 84000222 - Great Plains Health - Nephrology, North Platte, Nebraska
  - 84000420 - DaVita Clinical Research - Henderson, Henderson, Nevada
  - 84000337 - Kidney Specialists of Southern Nevada, Las Vegas, Nevada
  - 84000148 - Sierra Nevada Specialty Care, Reno, Nevada
  - 84000141 - Seacoast Kidney and Hypertension Specialists, Portsmouth, New Hampshire
  - 84000436 - Hypertension & Nephrology Association, Eatontown, New Jersey
  - 84000452 - New Jersey Kidney Care, Jersey City, New Jersey
  - 84000184 - Mattoo & Bhat Medical Associates, P.C., College Point, New York
  - 84000393 - NYU Langone Hospital - Long Island, Mineola, New York
  - 84000155 - DaVita Clinic Research Bronx, The Bronx, New York
  - 84000276 - Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York
  - 84000191 - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - 84000150 - Durham Nephrology Associates, PA, Durham, North Carolina
  - 84000232 - East Carolina University, Greenville, North Carolina
  - 84000410 - North Carolina Nephrology, PA, Raleigh, North Carolina
  - Nephrology Associates of the Carolinas, Shelby, North Carolina
  - 84000548 - HNC Dialysis, Ltd., Columbus, Ohio
  - 84000234 - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - 84000192 - Columbia Nephrology, Columbia, South Carolina
  - 84000367 - Dialysis Clinic, Inc., Spartanburg, South Carolina
  - 84000229 - DaVita Clinical Research, Spartanburg, South Carolina
  - 84000547 - Southeast Renal Research Institute, Chattanooga, Tennessee
  - 84000361 - Dialysis Clinic Inc - University Nephology, Knoxville, Tennessee
  - 84000180 - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - 84000451 - Cussimanio Research Group LLC, Austin, Texas
  - 84000438 - Research Management, Inc., Austin, Texas
  - 84000549 - MW Clinical Research Center, Beaumont, Texas
  - Dallas V.A. Medical Center, Dallas, Texas
  - 84000457 - US Renal Care, Dallas, Texas
  - 84000354 - Davita Clinical Research, El Paso, Texas
  - 84000421 - DaVita Clinical Research - Horizon, El Paso, Texas
  - 84000458 - Fort Worth Renal Group, Fort Worth, Texas
  - 84000649 - Clinical Research Strategies, Houston, Texas
  - 84000350 - DaVita Clinical Research, Houston, Texas
  - 84000498 - DaVita Clinical Research, Houston, Texas
  - 84000598 - Aqua Research Institute, Houston, Texas
  - Gulf Coast Clinical Research, Houston, Texas
  - 84000450 - Houston Medical Research Institute, LLC, Houston, Texas
  - 84000360 - Clinical Research Strategies, Inc., Houston, Texas
  - 84000196 - Southwest Houston Research, Houston, Texas
  - 84000880 - Laguna Clinical Research Associates, LLC, Laredo, Texas
  - 84000634 - Prime Clinical Research, Inc., Mansfield, Texas
  - 84000373 - Gamma Medical Research, Inc., McAllen, Texas
  - 84000324 - National Institute of Clinical Research, Inc., San Antonio, Texas
  - 84000351 - DaVita Clinical Research, San Antonio, Texas
  - 84000419 - Davita Clinical Research, San Antonio, Texas
  - 84000553 - DCR-San Antonio Stone Oak, San Antonio, Texas
  - 84000339 - DaVita Clinical Research North Houston, Shenandoah, Texas
  - 84000660 - Medrasa Clinical Research, Sherman, Texas
  - 84000551 - Renal Research of Montgomery County, The Woodlands, Texas
  - 84000535 - DCR-Norfolk Great Bridge, Chesapeake, Virginia
  - 84000424 - Nephrology Associates of Northern Virginia Inc, Fairfax, Virginia
  - 84000138 - Peninsula Kidney Associates, Hampton, Virginia
  - 84000156 - Tidewater Kidney Specialists, Norfolk, Virginia
  - 84000336 - Nephrology and Hypertension Associates, Bluefield, West Virginia
- Argentina (5):
  - FME Lomas de Zamora, Banfield
  - FME Mansilla, Buenos Aires
  - FME Formosa, Formosa
  - Nextdial S.A., Mar del Plata
  - Fresenius Tucumán, San Miguel de Tucumán
- Australia (17):
  - 03600023 - Royal North Shore Hospital (RNSH), Saint Leonards, New South Wales
  - 03600017 - Concord Repatriation General Hospital, Sydney, New South Wales
  - 03600037 - Cairns Hospital, Cairns, Queensland
  - 03600021 - Sunshine Coast University Private Hospital, Nambour, Queensland
  - 03600014 - Princess Alexandra Hospital, Woolloongabba, Queensland
  - 03600013 - Monash Medical Centre, Clayton, Victoria
  - 03600011 - Sunshine Hospital, St Albans, Victoria
  - 03600056 - Wide Bay Hospital and Health Service, Bundaberg
  - 03600060 - Austin Hospital, Heidelberg
  - 03600050 - Fiona Stanley Hospital, Murdoch
  - 03600021 - Sunshine Coast University Private Hospital, Nambour
  - 03600041 - Royal Melbourne Hospital, Parkville
  - 03600020 - Gold Coast University Hospital, Southport
  - 03600038 - Fraser Coast Renal Service, Hervey Bay Hospital, Urraween
  - 03600058 - Sydney Adventist Hospital, Wahroonga
  - 03600012 - Westmead Hospital, Westmead
  - 03600048 - Wollongong Renal Unit, Wollongong
- 04000006 - Wiener Gesundheitsverbund - Klinik Hietzing, Vienna, Austria
- Belgium (10):
  - 05600011 - Onze-Lieve-Vrouwziekenhuis VZW, Aalst
  - 05600005 - Imelda Ziekenhuis, Bonheiden
  - Centre Hospitalier Universitaire (CHU) de Charleroi - Hopital Civil Marie Curie, Charleroi
  - 05600004 - AZ Sint-Lucas, Ghent
  - 05600013 - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - Jan Yperman Ziekenhuis, Leper
  - 05600012 - Universitair Ziekenhuis Leuven, Leuven
  - 05600003 - CHR de la Citadelle, Liège
  - 05600018 - AZ Delta (H.-Hartziekenhuis Roeselare-Menen vzw (HHRM)) - Campus Rumbeke, Roeselare
  - 05600014 - VITAZ, Department Nierziekten & Dialyse, Sint-Niklaas
- Brazil (2):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Fundacao Pro Rim de Santa Catarina, Joinville
- Bulgaria (11):
  - Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich
  - 10000004 - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Sykehuset Østfold Kalnes, Grålum
  - 10000002 - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz - LOM EOOD, Lom
  - 10000009 - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - 10000007 - UMHAT Plovdiv, Plovdiv
  - 10000011 - Multiprofile Hospital for Active Treatment Dr. Ivan Seliminski - Sliven AD, Sliven
  - 10000001 - Medical Center - Smolyan OOD, Smolyan
  - University Hospital for Active Treatment Tsaritsa Joanna ISUL EAD, Sofia
  - 10000005 - Dialysis Center VIA DIAL OOD, Stara Zagora
  - 10000008 - UMHAT Prof. Dr. Stoyan Kirkovich, Stara Zagora
- Canada (14):
  - 12400008 - University of Alberta Hospital, Edmonton, Alberta
  - 12400021 - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - 12400026 - St. Josephs Healthcare Hamilton, Hamilton, Ontario
  - 12400009 - Kingston Health Sciences Centre, Kingston, Ontario
  - 12400030 - London Health Sciences Centre - University Hospital, London, Ontario
  - 12400024 - Lakeridge Health Oshawa, Oshawa, Ontario
  - 12400023 - McGill University Health Centre, Montreal, Quebec
  - 12400015 - Hôpital du Sacré-Cœur-de-Montréal, Montreal, Quebec
  - 12400014 - Maisonneuve-Rosemont Hospital, Montreal
  - 12400031 - CHUM - Centre hospitalier de l'Universite de Montreal, Montreal
  - 12400048 - Ciussse-Chus, Sherbrooke
  - 12400032 - St. Michaels Hospital, Toronto
  - 12400016 - St Paul Hospital, Vancouver
  - 12400027 - Seven Oaks Hospital, Winnipeg
- China (27):
  - Inner Mongolia Baotou City Central Hospital (Baotou Central Hospital), Baotou Shi
  - 15600014 - Peking University First Hospital, Beijing
  - 15600036 - Beijing Tsinghua Chang Gung Hospital, Beijing
  - 15600053 - People's Hospital of Deyang, Deyang Shi
  - 15600033 - Anhui Medical University-The Second Hospital, Hefei
  - The First Hospital of Jiaxing, Jiaxing
  - 15600019 - Gansu Provincial People's Hospital, Lanzhou
  - Henan University of Science and Technology-The First Affiliated Hospital, Luoyang Shi
  - 15600045 - Nanchang University - The First Affiliated Hospital, Nanchang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - 15600052 - The People's Hospital Guangxi Zhuang of Autonomous Region, Nanning
  - 15600035 - Southern Medical University - Jiangxi Pingxiang People's Hospital, Pingxiang
  - 15600034 - Shanghai Jiao Tong University School of Medicine (SJTUSM)-Renji Hospital, Shanghai
  - 15600030 - Shanghai First People's Hospital, Shanghai Shi
  - 15600049 - Shijiazhuang People's Hospital, Shijiazhuang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - 15600038 - Second Hospital of Shanxi Medical University, Taiyuan
  - 15600044 - Tianjin People's Hospital, Tianjin
  - 15600037 - Huazhong University of Science and Technology - Tongji Medical College - The Central Hospital of Wuhan (Wuhan Second Hospital), Wuhan
  - 15600015 - Wuxi People's Hospital, Wuxi
  - 15600018 - Zhongshan Hospital Xiamen University, Xiamen
  - 15600040 - Yan'an University Xianyang Hospital, Xianyang
  - 15600029 - Xinxiang City First People's Hospital, Xinxiang
  - 15600022 - Northern Jiangsu People's Hospital, Yangzhou
  - 15600025 - Yibin Second People's Hospital, Yibin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - 15600026 - Affiliated Hospital of Jiangsu University, Zhenjiang
- Denmark (5):
  - 20800009 - Aalborg Universitetshospital, Aalborg
  - 20800010 - Herlev Hospital, Herlev
  - 20800008 - Gødstrup Hospital, Herning
  - 20800011 - Trail Nation: Nordsjællands Hospital, Hillerød
  - Trial Nation: Holbæk Sygehus, Holbæk
- France (17):
  - 25000011 - CHU Amiens - Nephrology Dialysi Transplantation Department, Amiens
  - 25000014 - CHU de Saint-Étienne - Hôpital Nord, Aura
  - 25000027 - Centre Hospitalier Regional Universitaire (CHRU) Brest - Hopital de la Cavale Blanche, Brest
  - 25000013 - CHU de Caen, Caen
  - 25000032 - Fondation Charles Mion AIDER Santé, Grabels
  - 25000026 - Hopital Prive La Louviere, Lille
  - 25000033 - CHU de Limoges, Limoges
  - Hopitaux Universitaires de Marseille, Marseille
  - 25000018 - Centre Hospitalier Universitaire Montpellier - Hôpital Lapeyronie, Montpellier
  - CHE de Nice - Pasteur Hospital, Nice
  - 25000020 - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes
  - 25000028 - Hopital Pitie-Salpetriere, Paris
  - 25000025 - AURA Paris - Plaisance, Paris
  - 25000019 - Centre Hospitalier Universitaire (CHU) de Reims - Hopital Maison Blanche, Reims
  - 25000016 - AURA St Quen Dialysis centre, Saint-Ouen
  - 25000029 - Hôpitaux Universitaires de Strasbourg - Hôpital Civil, Strasbourg
  - 25000012 - CHU Rangueil, Toulouse
- Germany (7):
  - 27600047 - Charite-Universitatsmedizin Berlin, Berlin
  - 27600041 - Nierenzentrum Bad König, Hessen
  - 27600039 - Westpfalz Klinikum GmbH, Kaiserslautern
  - 27600022 - UKSH - Universitatsklinik Schleswig-Holstein, Kiel
  - 27600021 - Kuratorium fuer Dialyse und Nierentransplantation e.V. - KfH-Nierenzentrum - St. Georg, Leipzig
  - 27600040 - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - 27600020 - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
- Greece (13):
  - 30000015 - University Hospital of Alexandroupolis, Alexandroupoli
  - 30000016 - General Hospital of Arta, Arta
  - 30000012 - University General Hospital of Heraklion, Crete
  - 30000004 - University General Hospital of Ioannina, Ioannina
  - 30000002 - General Hospital of Ioannina G. Hatzikosta, Ioannina
  - 30000014 - Nephrological Clinic University Hospital, University of Thessaly, Larissa
  - 30000013 - General Hospital of Ptolemaida, Ptolemaida
  - 30000008 - University Hospital of Patras, Rio
  - 30000003 - AHEPA Univ. Hospital, Medical School, Aristotle University of Thessaloniki, Thessaloniki
  - 30000005 - Aristotle University, Hippokration, Thessaloniki
  - 30000006 - General Hospital of Thessaloniki, Agios Pavlos, Thessaloniki
  - 30000009 - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - 30000011 - Nephrology Department G. Papanikolaou General Hospital, Thessaloniki
- Hungary (2):
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - 34800012 - B. Braun Avitum - 14. Dialízisközpont Kistarcs, Kistarcsa
- Israel (7):
  - 37600008 - Carmel Medical Center, Haifa
  - 37600012 - Edith Wolfson Medical Center, Holon
  - 37600010 - Rabin Medical Center, Petah Tikva
  - 37600011 - Chaim Sheba Medical Center (Sheba Tel-Hashomer Medical Center ), Ramat Gan
  - 37600013 - Ziv Medical Center, Safed
  - 37600009 - Ichilov Hospital-Tel-Aviv Sourasky Medical Center, Tel Aviv
  - 37600002 - Medical Research & Development Fund for Health Services, PORIYA Hospital, Tiberias
- Italy (21):
  - 38000025 - ASST degli Spedali Civili di Brescia, Brescia
  - 38000031 - Azienda Ospedaliera Sant'Anna e San Sebastiano di Caserta, Caserta
  - 38000034 - AOU Policlinico G Rodolico - San Marco - Presidio Ospedaliero ospedale San Marco, Catania
  - 38000061 - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Ferrara
  - 38000074 - Ospedale Santa Maria Annunziata, Florence
  - 38000027 - A. O. -Universitaria Ospedali Riuniti di Foggia Farmacia Osp, Foggia
  - 38000059 - IRCCS Az. Osp. Universitaria San Martino- IST, Genova
  - 38000063 - Vito Fazzi Hospital in Lecce, Lecce
  - 38000024 - ASST di Lecco - Presidio Ospedaliero A. Manzoni di Lecco, Lecco
  - 38000029 - Università degli Studi di Messina, Messina
  - 38000017 - ASST Santi Paolo e Carlo - Ospedale San Carlo Borromeo, Milan
  - 38000023 - IRCCS Ospedale San Raffaele, Milan
  - 38000069 - Ospedale Maggiore di Novara, Novara
  - 38000019 - ICS Maugeri S.p.A. SB; Università di Pavia; Fondazione Salvatore Maugeri IRCCS, Pavia
  - 38000026 - University of Verona, Peschiera del Garda
  - 38000064 - AUSL Piacenza Hospital-Unit Nephrology Dialysis, Dept of Medicine, Piacenza
  - 38000032 - Ospedale Santo Stefan, Prato
  - 38000060 - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - 38000067 - Rimini Hospital, Rimini
  - 38000016 - Ospedale Casa Sollievo della Sofferenza (CSS), San Giovanni Rotondo
  - 38000020 - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Japan (31):
  - 39200053 - Daiyukai Daiichi Hospital, Ichinomiya-shi, Aichi-ken
  - 39200044 - Juntendo University Urayasu Hospital, Urayasu-shi, Chiba
  - 39200046 - Steel Memorial Yawata Hospital, Kitakyushu-shi, Fukuoka
  - 39200048 - Maebashi Hirosegawa Clinic, Maebashi, Gunma
  - 39200049 - Joumou Ohashi Clinic, Maebashi, Gunma
  - 39200045 - Teine Urological Clinic, Sapporo, Hokkaido
  - 39200054 - Omi freai Hospital, Kusatsu-shi, Shiga
  - 39200027 - Tokyo Womens Med University, Shinjuku-Ku, Tokyo
  - 39200042 - Matsunami General Hospital, Hashima-gun
  - 39200041 - Ishikiriseiki Hospital, Higashiosaka-shi
  - NHO Hiroshimanishi Medical Center, Hiroshima
  - 39200055 - Miki Internal Medicine Urology Clinic, Hokkaido
  - 39200033 - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun
  - 39200043 - Ueyama Hospital, Kagoshima
  - 39200021 - Kurume University Hospital, Kurume
  - 39200038 - St. Mary's Hospital, Kurume-shi
  - 39200028 - Rakuwakai Otowa Kinen Hospital, Kyoto
  - Matsubara Tokushukai Hospital, Matsubara-shi
  - 39200037 - Nagaoka Red-Cross Hospital, Nagaoka-Shi
  - 39200020 - Chubu Rosai Hospital, Nagoya
  - 39200035 - Daido Hospital, Nagoya
  - 39200032 - Oguranaika Jin Cinic, Oyama-shi
  - 39200026 - Omihachiman Community Medical Center - Kidney Center, Ōmihachiman
  - 39200029 - Ibaraki Seinan Medical Center Hospital, Sakaimachi
  - 39200031 - Kurosawa Hospital, Takasaki-Shi
  - Centrul Medical de Nefrologie si Dializa Diaverum Targu Mures, Târgu Mureș
  - 39200034 - Kikuchi Medical Clinic, Tsukuba
  - 39200030 - St.Hill Hospital, Ube-shi
  - Yamagata Tokushukai Hospital, Yamagata
  - 39200051 - Bosei Kannai Clinic, Yokohama
  - 39200036 - Sanin Rosai Hospital, Yonago-shi
- Malaysia (3):
  - Hospital Raja Permaisuri Bainun, Ipoh, Ipoh
  - Queen Elizabeth Hospital, Kota Kinabalu
  - Seberang Jaya Hospital, Perai
- Norway (2):
  - 57800004 - Vestre Viken HF - Drammen Sykehus (Sykehuset Buskerud), Drammen
  - Sykehuset Telemark, Skien
- Poland (4):
  - Davita Stacja Dializ w Brodnicy, Brodnica
  - 61600011 - Powiatowy Szpital Specjalistyczny w Stalowej Woli, Stalowa Wola
  - 61600022 - Diaverum - NZOZ Tczewie, Tczew
  - 61600025 - DaVita Stacja Dializ, Warsaw
- Portugal (7):
  - 62000011 - Unidade Local de Saúde de Braga, E. P. E., Braga
  - NephroCare Carregado, Carregado
  - Centro Hospitalar e Universitário de Lisboa Centra, Lisbon
  - 62000010 - Unidade Local de Saúde de Loures -Odivelas, E. P. E., Loures
  - 62000009 - Unidade Local de Saúde de São José, E. P. E., Oeiras
  - 62000005 - Unidade Local de Saúde de Santo António, E. P. E., Porto
  - 62000007 - Unidade Local de Saúde do Estuário do Tejo, E. P. E., Vila Franca de Xira
- Romania (14):
  - Centrul de Dializa Fresenius NephroCare Brasov, Brasov
  - 64200014 - SC International Healthcare Systems SA - IHS Sf. Ioan Dialysis Center, Bucharest
  - Centrul de Dializa Fresenius NephroCare Bucaresti, Bucharest
  - 64200024 - Fundeni Clinical Institute, Bucharest
  - Centrul de Nefrologie si Dializa DIAVERUM Sema Parc, Bucharest
  - Centrul de Nefrologie si Dializa Diaverum Fundeni, Bucharest
  - Centrul de Dializa Fresenius NephroCare Cluj, Cluj-Napoca
  - Centrul de Dializa Fresenius NephroCare Constanta, Constanța
  - 64200016 - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Constanta (Emergency Clinic Hospital Constanta), Constanța
  - Centrul de Nefrologie si Dializa Diaverum Craiova, Craiova
  - 64200026 - Spitalul Clinic -Dr. C.I. Parhon - Iasi, Iași
  - Spitalul Clinic Municipal Dr. Gavril Curteanu Oradea, Oradea
  - Centrul de Dializa Fresenius NephroCare Ploiesti, Ploieşti
  - 64200005 - Spital Judetean de Urgenta Satu Mare, Satu Mare
- Slovakia (2):
  - 70300002 - LC-REN s.r.o., Lučenec
  - Biodial, s.r.o., Púchov
- South Korea (10):
  - 41000002 - SMG - SNU Boramae Medical Center, Ilsan-gu, Seoul
  - 41000006 - Hallym University Sacred Heart Hospital, Anyang-si
  - 41000004 - Keimyung University Dongsan Medical Center, Daegu
  - 41000001 - Gangnam Severance Hospital, Gangnam-gu
  - 41000009 - National Health Insurance Service - Ilsan Hospital, Goyang-si
  - 41000010 - Hanyang University Guri Hospital, Guri-si
  - 41000008 - Konkuk University Medical Center, Gwangju
  - 41000005 - Seoul National University Hospital, Seoul
  - 41000012 - Severance Hospital, Yonsei University, Seoul
  - 41000007 - Yonsei University - Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - Centro de dialisis Alcobendas, Alcobendas
  - Hospital Universitario Valle de Hebron, Barcelona
  - 72400019 - Hospital Universitari de Girona Dr Josep Trueta, (Avitum), Girona
  - 72400011 - Universidad de Alcala (UAH), Guadalajara
  - 72400007 - Hospital Universitari Arnau de Vilanova, Lleida
  - 72400012 - Hospital de Manises, Manises
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela
  - 72400031 - Hospital Clinico Universitario - Valencia, Valencia
  - 72400008 - Hospital Universitari i Politècnic La Fe, Valencia
- 75200001 - Uppsala Universitet - Akademiska Sjukhuset, Uppsala, Sweden
- United Kingdom (15):
  - 82600041 - University Hospitals Birmingham NHS Foundation Trust - Birmingham Heartlands Hospital (BHH), Birmingham
  - 82600027 - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - 82600023 - University Hospital Coventry and Warwickshire, Coventry
  - 82600060 - University Hospitals of Derby and Burton NHS Foundation Trust - Royal Derby Hospital, Derby
  - 82600022 - Dorset County Hospital NHS Foundation Trust - Dorset County Hospital (DCH), Dorchester
  - 82600024 - Royal Liverpool University Hospital, Liverpool
  - 82600026 - William Harvey Research Institute ; Barts Health NHS Trust - The Royal London Hospital, London
  - 82600032 - King´s College NHS Trust, London
  - 82600034 - St George's University Hospitals NHS Foundation Trust - St G, London
  - 82600042 - Hammersmith Hospital Imperial College Healthcare NHS Trust -Hammersmith Hospital - West London Renal and Transplant Centre, London
  - 82600028 - Altnagelvin Area Hospital, Londonderry
  - 82600029 - Northern Care Alliance NHS Foundation Trust - Salford Royal NHS Foundation Trust-Salford Care Organisation, Salford
  - 82600039 - The Shrewsbury and Telford Hospital NHS Trust (SaTH) - Royal Shrewsbury Hospital, Shrewsbury
  - 82600025 - Royal Stoke University Hospital, Stoke-on-Trent
  - 82600049 - The Royal Wolverhampton NHS Trust - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

REFERENCES:
- [Derived] Chertow GM, Chang AM, Felker GM, Heise M, Velkoska E, Fellstrom B, Charytan DM, Clementi R, Gibson CM, Goodman SG, Jardine M, Levin A, Lokhnygina Y, Mears J, Mehran R, Stenvinkel P, Wang AY, Wheeler DC, Zoccali C, Ridker PM, Mahaffey KW, Tricoci P, Wolf M. IL-6 inhibition with clazakizumab in patients receiving maintenance dialysis: a randomized phase 2b trial. Nat Med. 2024 Aug;30(8):2328-2336. doi: 10.1038/s41591-024-03043-1. Epub 2024 May 25. PMID 38796655